CLINICAL TRIAL: NCT02655978
Title: Rostral Dorsal Cingulum Bundle Connectivity in Patients With Bipolar Disorder
Status: Completed | Type: Observational
Sponsor: University Hospitals Cleveland Medical Center (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Principal Investigator, Jennifer Sweet, MD, Neurosurgeon, University Hospitals Cleveland Medical Center
Other Study IDs: 02-15-35; KL2TR000440 (NIH)
Record Dates: First submitted 2016-01-06; First posted 2016-01-14 (Estimated); Last update posted 2020-11-12 (Actual); Status verified 2020-11

CONDITIONS: Bipolar Disorder
MeSH Terms: conditions — Bipolar Disorder | interventions — Magnetic Resonance Spectroscopy

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Healthy Volunteers: These participants will not have any psychiatric disorder as assessed by a structured clinical interview for psychiatric disorders.
  Interventions: Other: Magnetic Resonance Imaging
- Medically Treatment-Responsive BD: This group will be composed of participants who have BDI or BDII and have most recently been depressed but are currently in remission with evidence-based treatments for bipolar disorder
  Interventions: Other: Magnetic Resonance Imaging
- Treatment-Refractory BD: This group will be composed of participants who have BDI or BDII, are currently depressed with their current episode lasting at least 12 months and not responding to 4 adequate evidence-based treatments for BDI or BDII and who have failed, been intolerant to, or were unwilling to try electroconvulsive therapy (ECT).
  Interventions: Other: Magnetic Resonance Imaging

INTERVENTIONS:
Other: Magnetic Resonance Imaging

SUMMARY:
The overall goal of this study is to employ diffusion-weighted imaging (DWI) and tractography to investigate differences in connectivity in the rostral dorsal cingulum bundle (CB) in patients with bipolar disorder type I (BDI) or bipolar type II (BDII) compared to matched controls, and to utilize this information to determine if high-frequency deep brain stimulation (DBS) of the rostral dorsal CB has realistic potential as a therapy for producing mood stabilization in patients with BDI or BDII.

ELIGIBILITY:
1. Inclusion and Exclusion Criteria for Group 1: Healthy Volunteers

   a. Inclusion Criteria for Group 1:

   i. Male or female, age 18 or older

   ii. In the opinion of the investigator, capable of understanding and complying with protocol requirements

   iii. In the opinion of the investigator, has the competency to understand and sign the informed consent

   iv. Physically healthy

   v. Without any current and/or lifetime psychiatric disorder assessed with a Structured Clinical Interview for psychiatric Disorders, including the Mini International Neuropsychiatric Interview (MINI)

   b. Exclusion Criteria for Group 1:

   i. Significant structural brain lesion identified (e.g. infarct, hemorrhage, tumor, multiple sclerosis)

   ii. Progressive neurological disease such as neurodegenerative disease

   iii. Preexisting implanted electrical device (such as pacemaker or cardiac defibrillator)

   iv. Any psychiatric disorder including any severe personality disorder

   v. Currently pregnant or planning to become pregnant

   vi. Any other contraindications to the brain imaging procedures.

   vii. Tests positive for illegal substances or prescription medications for which they do not have a valid prescription

   viii. Currently taking any steroids, stimulants, or opioid pain killers.

   ix. Currently experiencing nicotine dependence or any smoking of cigarettes or use of other nicotine containing products within a week before the imaging visit.
2. Inclusion and Exclusion Criteria for Group 2: Medically Treatment-Responsive Bipolar Disorder

   a. Inclusion Criteria for Group 2:

   i. Male or female, age 18 or older

   ii. In the opinion of the investigator, capable of understanding and complying with protocol requirements

   iii. In the opinion of the investigator, has the competency to understand and sign the informed consent

   iv. Meets diagnostic criteria for BDI or BDII according to the DSM-V criteria, as confirmed by a systematic clinical interview and the administration of the MINI

   v. A recent episode of depression, currently in remission with evidence-based treatments for bipolar disorder

   vi. Montgomery-Asberg Depression Rating Scale (MADRS) total score ≤ 10

   vii. Young Mania Rating Scale (YMRS, Young et al 1988) total score ≤ 8

   viii. Global Clinical Impression-Severity for Bipolar Disorder (CGI-S-BD) ≤ 2

   ix. Subject is compliant with taking medication per the investigator's discretion

   b. Exclusion Criteria for Group 2:

   i. Significant structural brain lesion identified (e.g. infarct, hemorrhage, tumor, multiple sclerosis)

   ii. Progressive neurological disease such as neurodegenerative disease

   iii. Preexisting implanted electrical device (such as pacemaker or cardiac defibrillator)

   iv. Contribution of any co-occurring psychiatric comorbidity that is disproportionate to the contribution of BDI or BDII, such as severe obsessive-compulsive disorder (OCD) or post-traumatic stress disorder (PTSD)

   v. Meets criteria for antisocial personality disorder

   vi. Meets criteria for having borderline personality disorder

   vii. There will be no exclusions based on prescribed CNS-active medications

   viii. Tests positive for illegal substances or prescription medications for which they do not have a valid prescription

   ix. Meets DSM-V criteria for any alcohol and/or drug use disorder within the last 6 months, excluding the use of caffeine and/or nicotine

   x. Currently pregnant or planning to become pregnant

   xi. Any other contraindications to the brain imaging procedures.
3. Inclusion and Exclusion Criteria for Group 3: Treatment-Refractory Bipolar Disorder

   a. Inclusion Criteria for Group 3:

   i. Male or female, age 18 or older

   ii. In the opinion of the investigator, capable of understanding and complying with protocol requirements

   iii. In the opinion of the investigator, has the competency to understand and sign the informed consent

   iv. Meets diagnostic criteria for BDI or BDII, currently depressed, at least moderately severe with or without psychotic features, according to the DSM-V criteria, as confirmed by a systematic clinical interview and the administration of the Structured Clinical Interview for Psychiatric Disorders, including the Mini International Neuropsychiatric Interview (MINI)

   v. Current episode lasting at least 6 months and not responding to 2 adequate evidence-based treatments for BDI or BDII assessed with the assistance of Modified Antidepressant Treatment History Form (MATHF) and verified through medical records if possible

   vi. If a subject has refused treatment with a particular FDA-approved mood stabilizer due to reasons of unacceptable side effects (such as weight gain, etc.), their wishes will be respected

   vii. Depression severity should be measured with Montgomery-Asberg Depression Rating Scale (MADRS). A MADRS total score ≥ 20 is required at Screening Visit/Baseline Evaluation.

   viii. Has experienced marked impairment as documented by a score consistent with severe impairment (7 or more on at least one of the three subscales of the Sheehan Disability Scale (SDS), which includes an assessment of work-life, family-life, and social life (no/mild impairment 0-3, moderate impairment 4-6, severe impairment 7-10)

   ix. Bipolar disorder and current depressive episode as the primary source of the patient's disability, according to both the subject and the psychiatrist

   b. Exclusion Criteria for Group 3:

   i. Significant structural brain lesion identified (e.g. infarct, hemorrhage, tumor, multiple sclerosis)

   ii. Progressive neurological disease such as neurodegenerative disease

   iii. Preexisting implanted electrical device (such as pacemaker or cardiac defibrillator)

   iv. Contribution of any co-occurring psychiatric comorbidity that disproportionate to the contribution of BDI or BDII, such as severe obsessive-compulsive disorder (OCD) or post-traumatic stress disorder (PTSD)

   v. Meets criteria for antisocial personality disorder

   vi. Meets criteria for having borderline personality disorder

   vii. There will be no exclusions based on prescribed CNS-active medications

   viii. Tests positive for illegal substances or prescription medications for which they do not have a valid prescription

   ix. Meets DSM-V criteria for any alcohol and/or drug use disorder within the last 6 months, excluding the use of caffeine and/or nicotine

   x. Active suicidal ideation with a plan or intent, a suicide attempt within past 6 months or more than 2 suicide attempts within the past 2 years

   xi. Currently pregnant or planning to become pregnant

   xii. Any other contraindications to the brain imaging procedures.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Participants from all three groups will be made up of those who respond to IRB approved advertisements or are referred by a provider within the UHCMC Department of Psychiatry or other provider referral.
Sampling Method: Non-Probability Sample
Enrollment: 45 (Actual)
Dates: Start 2016-01 (Actual); Primary Completion 2019-10 (Actual); Study Completion 2019-10 (Actual)

PRIMARY OUTCOMES:
Differences in connectivity in the rostral dorsal CB in patients with BDI or or BDII compared to matched controls | Day 1
  The imaging visit will consist of an MRI with diffusion-weighted imaging (DWI) sequences

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer A Sweet, MD, Principal Investigator — University Hospitals Cleveland Medical Center
Locations (1):
- University Hospitals Cleveland Medical Center, Cleveland, Ohio, United States